CLINICAL TRIAL: NCT02977312
Title: Observational Study of Cemivil® (Imatinib) in Chronic Myeloid Leukemia Patients in Jordan
Brief Title: Study of Cemivil® (Imatinib) in Chronic Myeloid Leukemia Patients in Jordan
Acronym: CCMLJ
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Cemivil-2011-01
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Imatinib — Observation of chronic myeloid leukemia (CML) patients in chronic phase (CP) treated with Cemivil
  Other Names: Cemivil

SUMMARY:
This study assessed the efficacy and safety of generic imatinib in patients with chronic myeloid leukemia (CML) in Jordan. It was a multicenter, non-interventional, open-label, prospective study combined with retrospective data collection from files of patients with a diagnosis of Ph+ CML, treated with Cemivil (imatinib), where no visits or intervention(s) additional to the daily practice were performed

DETAILED DESCRIPTION:
Primary objectives

Measure the proportion of Philadelphia chromosome positive (Ph+) CML patients in CP treated with Cemivil who achieve optimal response :

* Complete hematologic response (CHR) at 3 months;
* Minor cytogenetic response (mCyR) at 3 months (Ph+ ≤65%); partial cytogenetic response (PCyR) at 6 months (Ph+ ≤35%), and complete cytogenetic response (CCyR) at 12 months (No Ph+ metaphases);
* Major molecular response (MMR) at 12 months of Cemivil therapy [a ratio of BCR-ABL1 to ABL1 ≤0.1% on the International Scale];

Assess the safety and tolerability of Cemivil after one year of treatment, based on:

* Incidence, severity, and relationship of adverse events (AEs) to the study medication;
* Serious AEs;
* AEs leading to permanent treatment discontinuation;
* Clinically relevant changes in laboratory tests (according to laboratory reference ranges).

Number of Subjects evaluated: 91 (N=33 received generic imatinib as first-line therapy "first-line patients". N=58 switched from patented imatinib to generic imatinib "switched patients")

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Newly diagnosed patients with Ph+ CML in CP; or CML patients who started with Cemivil treatment since its registration in Jordan and who confirmed CHR
* Written informed consent

Exclusion Criteria:

* Age <18 years
* CML in accelerated phase
* CML in blast crisis
* CML with mutation(s) in the BCR-ABL gene
* Contraindications to the administration of the study drug according to the approved Summary of Product Characteristics (SPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) patients in chronic phase (CP)
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rate of Complete Cytogenetic Response (CCyR) | 12 months
Rate of Major Molecular Response (MMR) | 12 months

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | 12 months
  (Safety & Tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Abbadi, Professor, Principal Investigator — Jordan University Hospital
Locations (3):
- Jordan (3):
  - Al Bashir Hospital, Amman
  - Jordan University Hospital, Amman
  - King Hussein Cancer Center, Amman

IPD SHARING:
Plan to Share IPD: No